CLINICAL TRIAL: NCT02088892
Title: A Clinical Challenge Study to Quantify BCG at the Challenge Site of Healthy Volunteers Receiving Either Intradermal BCG SSI or BCG TICE at Standard or High Dose
Brief Title: A Clinical Challenge Study of BCG in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Aeras (Other); University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: TB031
Record Dates: First submitted 2014-03-10; First posted 2014-03-17 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Tuberculosis
Keywords: BCG challenge study
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Experimental): 10 BCG-naïve subjects receiving intradermal BCG SSI at standard dose (2-8 x 10^5 cfu) followed by a punch biopsy at the challenge site 14 days later.
  Interventions: Drug: BCG SSI
- Group B (Experimental): 10 BCG-naïve subjects receiving BCG Tice at standard dose (2-8 x 10^5 cfu) followed by a punch biopsy at the challenge site 14 days later.
  Interventions: Drug: BCG Tice
- Group C (Experimental): 10 BCG-naïve subjects receiving intradermal BCG SSI at high dose (6-24 x 10^5 cfu) followed by a punch biopsy at the challenge site 14 days later.
  Interventions: Drug: BCG SSI
- Group D (Experimental): 10 BCG-naïve subjects receiving intradermal BCG Tice at high dose (6-24 x 10^5 cfu) followed by a punch biopsy at the challenge site 14 days later.
  Interventions: Drug: BCG Tice
- Group E (Experimental): 8-12 BCG-naïve subjects receiving the optimal strain and dose of intradermal BCG identified from preliminary results obtained from Group A, B, C and D, followed by a punch biopsy at the challenge site 14 days later.
  Interventions: Drug: BCG SSI; Drug: BCG Tice

INTERVENTIONS:
Drug: BCG SSI — Intradermal injection
  Other Names: Bacille Calmette-Guérin Statens Serum Institute (BCG SSI)
  Arms: Group A; Group C; Group E
Drug: BCG Tice — Intradermal injection
  Other Names: Bacille Calmette-Guérin Tice
  Arms: Group B; Group D; Group E

SUMMARY:
TB031 is a challenge study comparing two different strains of the Bacille Calmette-Guérin (BCG) vaccine at standard and high dose.

DETAILED DESCRIPTION:
Currently, to assess vaccine efficacy against tuberculosis (TB) there is no alternative to large randomized controlled trials. These efficacy trials for novel TB vaccines are difficult, long and very costly. For this reason there is an urgent need for a valid, reliable, and strong correlate of protection which can help distinguish between candidate TB vaccines undergoing phase I trials, and thereby allow the vaccine development field to advance more quickly, and in a more cost-effective manner.

This study aims to address the current lack of immunological correlates in the TB vaccine field. As an alternative to phase II field trials, human challenge models can provide an evaluation of preliminary efficacy of vaccine candidates. Challenge models, with their concept of deliberate infectious challenge of human volunteers, have been well established for pathogens such as malaria, typhoid and dengue, and these models have greatly facilitated vaccine development. At present there is no safe human challenge model of Mycobacterium tuberculosis (M. tb) infection to enable proof-of-concept efficacy evaluation of candidate vaccines.

Whilst scientists cannot use M. tb as a challenge agent to evaluate efficacy in a clinical trial for safety and ethical reasons, they can use another mycobacterium, attenuated Mycobacterium bovis, as a surrogate for M. tb infection. Attenuated Mycobacterium bovis is the mycobacterial strain in BCG and is safe to use in humans. An effective vaccine against M. tb should also be effective against BCG. After injection into humans, BCG replicates, and an effective TB vaccine should reduce this BCG replication. The BCG challenge model is based on this premise. In the human BCG challenge model, BCG is administered intradermally and the degree of BCG growth suppression is quantified by analysing the tissue obtained in a punch biopsy of volunteers' skin over the BCG 'challenge' site.

This study aims to use two different strains of BCG, each at standard and high dose, to optimise this BCG challenge model.

ELIGIBILITY:
Inclusion Criteria:

Volunteers must meet all of the following criteria to enter the study:

* Healthy adult aged 18-55 years
* BCG naïve
* Resident in or near Oxford (for CCTVM) or Birmingham (for WTCRF) for the duration of the study period
* No relevant findings in medical history or on physical examination
* Allow the Investigators to discuss the volunteer's medical history with their GP
* Use effective contraception for the duration of the study period (females only)
* Agreement to refrain from blood donation during the duration of the study
* Give written informed consent
* Allow the Investigator to register volunteer details with a confidential database to prevent concurrent entry into clinical trials
* Able and willing (in the Investigator's opinion) to comply with all the study requirements

Exclusion Criteria:

Volunteers must meet none of the following criteria to enter the study:

* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Previous vaccination with BCG, or any candidate TB vaccine
* Within the last year had close household contact with an individual with smear positive pulmonary tuberculosis
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* History of serious psychiatric condition
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the challenge agent
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the study
* Positive HBsAg, HCV or HIV antibodies
* Female confirmed pregnant or intention to become pregnant during study period, or currently lactating
* Current involvement in another trial that involves regular blood tests or an investigational medicinal product
* Use of an investigational medicinal product or non-registered drug, live vaccine, or investigational medical device for four weeks prior to dosing with the study challenge agent
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned challenge date
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk, or may influence the result of the study, or may affect the volunteer's ability to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Quantity of BCG at challenge site | At Day 14
  To evaluate and compare the amount of BCG (measured by CFU count and PCR) from a biopsy taken from the intradermal BCG challenge site in healthy BCG-naïve adults receiving either BCG SSI or BCG Tice at either standard or high dose

SECONDARY OUTCOMES:
Immune response markers | Up to Day 14
  To identify laboratory markers of the immune response that correlate with the levels of mycobacterial suppression at the BCG challenge site

OTHER OUTCOMES:
Local and systemic adverse events | Up to Day 28
  To evaluate and compare local and systemic adverse events between the different challenge models through actively and passively collected data on adverse events.
Mycobacterial Growth Inhibition Assays | Up to day 14
  Use of Mycobacterial Growth Inhibition Assays to evaluate the effect of recent BCG vaccination on in-vitro ability to control Staphylococcus aureus, and potentially also Klebsiella, Group B streptococcus and Escherichia coli.

CONTACTS AND LOCATIONS:
Overall Officials: Helen McShane, Study Director — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine, University of Oxford, Oxford, Oxfordshire
  - The Wellcome Trust Clinical Research Facility, University of Birmingham, Birmingham, West Midlands

REFERENCES:
- [Derived] Minhinnick A, Harris S, Wilkie M, Peter J, Stockdale L, Manjaly-Thomas ZR, Vermaak S, Satti I, Moss P, McShane H. Optimization of a Human Bacille Calmette-Guerin Challenge Model: A Tool to Evaluate Antimycobacterial Immunity. J Infect Dis. 2016 Mar 1;213(5):824-30. doi: 10.1093/infdis/jiv482. Epub 2015 Oct 8. PMID 26450421
- See also: Jenner Institute Clinical Trials — http://www.jenner.ac.uk/clinicaltrials